CLINICAL TRIAL: NCT05052853
Title: Early Intervention of Prodromal Schizophrenia Using an NMDA Enhancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMUH110-REC3-114
Record Dates: First submitted 2021-09-08; First posted 2021-09-22 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Prodromal Schizophrenia
Keywords: Schizophrenia; Prodrome; NMDA
MeSH Terms: conditions — Schizotypal Personality Disorder; Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NMDAE (Experimental): An NMDA enhancer
  Interventions: Drug: NMDAE
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo Cap

INTERVENTIONS:
Drug: NMDAE — Use of an NMDA enhancer for the treatment of prodromal schizophrenia .
  Arms: NMDAE
Drug: Placebo Cap — Use of placebo as a comparator
  Arms: Placebo

SUMMARY:
Previous studies found that some NMDA-enhancing agents were able to improve clinical symptoms of patients with schizophrenia. Whether treatment of an NMDA-enhancing agent can benefit the treatment of prodromal schizophrenia deserves study.

DETAILED DESCRIPTION:
Several lines of evidence suggest that NMDA hypotheses have been implicated in schizophrenia. Previous studies found that some NMDA-enhancing agents were able to benefit the treatment of schizophrenia. Whether an NMDA-enhancer (NMDAE) can benefit the treatment of prodromal schizophrenia deserves study. Therefore, this study aims to compare NMDAE and placebo in the treatment of prodromal schizophrenia.

The subjects with prodromal schizophrenia at first receive 6 weeks of health-promotion intervention (including exercise and education). A total of 48 subjects who do not respond sufficiently to the health-promotion program are then recruited to this 12-week, randomized, double-blind, placebo-controlled trial, which aims to compare treatment response of NMDAE vs. placebo in 1:1 ratio. Clinical performances and side effects are measured at weeks -6 (before the screening phase), 0 (baseline of the drug trial), 2, 4, 6, 9, and 12. Cognitive functions are assessed at baseline and at endpoint of treatment by a battery of tests.

The efficacies of NMDAE and placebo will be compared. Chi-square (or Fisher's exact test) will be used to compare differences of categorical variables and t-test (or Mann-Whitney test if the distribution is not normal) for continuous variables between treatment groups. Mean changes from baseline in repeated-measure assessments will be assessed using the generalized estimating equation (GEE). All p values for clinical measures will be based on two-tailed tests with a significance level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Individuals meeting Criteria of Prodromal Syndrome (at least one of the following: 1. attenuated positive symptoms; 2. brief intermittent psychotic symptoms; 3. genetic risk and deterioration).
* Subjects remain symptomatic (scoring at least 20 on the Scale of Prodromal Symptoms [SOPS] total score) after the 6-week screening phase (which contains the health-promotion program) and before the 12-week drug-trial period.
* Subjects may be receiving ongoing treatment with antipsychotic medications, or may be medication-free for at least 12 weeks.For the subjects who have already been on such medications, the medications need to be continued for at least 4 weeks before the screening phase and the doses need to be kept unchanged during the study period. For those who have not yet been on such medications, these medications are forbidden during the study period.
* Subjects agree to participate in the study and provide written informed consent after complete description of the study. For the subject < 20 years old, a parent also has to provide written informed consent.

Exclusion Criteria:

* DSM-5 diagnosis of intellectual disability, substance (including alcohol) use disorder, schizophrenia, schizophreniform disorder, delusional disorder, schizoaffective disorder, substance/medication-induced psychotic disorder, or psychotic disorder due to another medical condition.
* History of epilepsy, head trauma, stroke, or serious medical or central nervous system diseases (other than schizophrenia) which may interfere with the study.
* Clinically significant laboratory screening tests (including blood routine, biochemical tests)
* Pregnancy or lactation
* Inability to follow protocol

Ages: 13 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Scale of Prodromal Symptoms [SOPS] total score | week 0, 2, 4, 6, 9, 12
  Assessment of overall prodromal symptoms. Minimum value: 0, maximum value: 114, the higher scores mean a worse outcome.
  As shown in "Detailed Description", "mean changes from baseline in repeated-measure assessments will be assessed using the generalized estimating equation (GEE). That is, GEE is used for analyzing the changes from baseline in repeated-measure assessments by a single analysis (but not multiple analyses).

SECONDARY OUTCOMES:
Change from baseline in SOPS Positive Symptom Scale score | week 0, 2, 4, 6, 9, 12
  Assessment of positive prodromal symptoms. Minimum value: 0, maximum value: 30, the higher scores mean a worse outcome.
Change from baseline in SOPS Negative Symptom Scale score | week 0, 2, 4, 6, 9, 12
  Assessment of negative prodromal symptoms. Minimum value: 0, maximum value: 36, the higher scores mean a worse outcome.
Change from baseline in SOPS Disorganization Symptom Scale score | week 0, 2, 4, 6, 9, 12
  Assessment of disorganization prodromal symptoms. Minimum value: 0, maximum value: 24, the higher scores mean a worse outcome.
Change from baseline in SOPS General Symptom Scale score | week 0, 2, 4, 6, 9, 12
  Assessment of general prodromal symptoms. Minimum value: 0, maximum value: 24, the higher scores mean a worse outcome.
Change from baseline in Scales for the Assessment of Negative Symptoms (SANS) total score | week 0, 2, 4, 6, 9, 12
  Assessment of schizophrenia negative symptoms. Minimum value: 0, maximum value:100, the higher scores mean a worse outcome.
Change from baseline in Clinical Global Impression | week 0, 2, 4, 6, 9, 12
  Assessment of general impression. Minimum value: 1, maximum value:7, the higher scores mean a worse outcome.
Change from baseline in Global Assessment of Functioning | week 0, 2, 4, 6, 9, 12
  Assessment of social, occupational, and psychological function. Minimum value: 1, maximum value:100, the higher scores mean better function.
Change from baseline in Hamilton Rating Scale for Depression | week 0, 2, 4, 6, 9, 12
  Assessment of depressive symptoms. Minimum value: 0, maximum value:52, the higher scores mean a worse outcome.
Change from baseline in Quality of Life Scale | week 0, 2, 4, 6, 9, 12
  Assessment of life quality. Minimum value: 0, maximum value:126, the higher scores mean a better outcome.
Change from baseline in Cognitive function | Week 0, 12
  The measure is the composite from multiple measures. All tests have no unit. For the domain (a. and c.) with more than one test, a composite T score will be calculated by standardizing the average of each T score. Furthermore, a global composite score (for all seven domains) and a neurocognitive composite score (for the first 6 domains, a-f) will be also calculated by standardizing the average of the T score of each domain (Lane HY et al, JAMA Psychiatry. 2013).
  Ten tests for assessment of 7 cognitive domains:
  1. speed of processing (assessed by Category Fluency, Trail Marking A, WAIS-III Digit Symbol-Coding);
  2. sustained attention (Continuous Performance Test);
  3. working memory: verbal (digit span) and nonverbal (spatial span);
  4. verbal learning and memory (WMS-III, word listing);
  5. visual learning and memory (WMS-III, visual reproduction);
  6. reasoning and problem solving (WISC-III, Maze);
  7. social cognition (MSCEIT Version 2)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, China Medical University Hospital, Taichung, Taiwan